CLINICAL TRIAL: NCT04000217
Title: A Randomized Control Trial Comparing Written Versus Verbal Brief Cognitive Behavioral Exposure Therapy Delivered Online
Brief Title: Written Versus Verbal Brief Cognitive Behavioral Exposure Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Responsible Party: Principal Investigator, Carmen McLean, Principal Investigator, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 640C89370
Record Dates: First submitted 2019-06-24; First posted 2019-06-27 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Written Exposure Therapy; Imaginal Exposure Therapy
MeSH Terms: interventions — Implosive Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Written Exposure Therapy (Active Comparator): Written exposure therapy (Sloan et al., 2012) is a brief evidence-based treatment for PTSD (US Dept. of VA & DoD, 2017), wherein patients are asked to write about their trauma memories for 30 minutes, with therapist instruction and feedback before and after each writing exercise.
  Interventions: Behavioral: Written Exposure Therapy
- Imaginal Exposure Therapy (Active Comparator): Imaginal exposure therapy will involve verbal recounting of trauma memories for 30 minutes with therapist instruction and feedback before and after each recounting exercise.
  Interventions: Behavioral: Imaginal Exposure Therapy

INTERVENTIONS:
Behavioral: Written Exposure Therapy — In this study, written exposure therapy is delivered in an online format with coaching from trained peer support specialists. Participants will complete 4-8 sessions, depending on their level of symptom reduction (i.e., allow for early termination when low symptom levels are achieved).
  Arms: Written Exposure Therapy
Behavioral: Imaginal Exposure Therapy — Delivery of imaginal exposure in this study will mirror the procedures used in WET. It will be delivered in an online format with coaching from trained peer support specialists. Participants will complete 4-8 sessions, depending on their level of symptom reduction (i.e., allow for early termination when low symptom levels are achieved).
  Arms: Imaginal Exposure Therapy

SUMMARY:
The purpose of the study is to compare the efficacy of two different versions of a brief online exposure therapy program for PTSD: written versus verbal trauma narrative recounting in reducing PTSD symptom severity. Both treatments will be delivered through an interactive online program with coaching from a trained peer support specialist. Treatment will be a variable length, such that 4 to 8 sessions will be delivered, depending on each participants' rate of PTSD symptom recovery.

ELIGIBILITY:
Inclusion Criteria:

* Able to read/write English
* Internet connection allowing stable access to the Vets Prevail website
* A clinically significant PCL-5 score of 31 or above.

Exclusion Criteria:

* A score on the suicidality item of the PHQ-9 of 3 or higher.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Post Traumatic Stress Disorder CheckList for Diagnostic and Statistical Manual - 5 (PCL-5; Weathers, et al., 2013) | Change in total score from baseline to 3-months post treatment (approximately 14-18 weeks).
  Self report measure of PTSD symptoms. A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items. Higher scores indicate greater PTSD severity.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9; Kroenke, Spitzer, & Williams, 2001). | Change in total score from baseline to 3-months post treatment (approximately 14-18 weeks).
  Self report measure of depression symptoms. It is the 9-item measure that yields a total score of 0-27, with higher scores indicating greater depressive symptom severity.
Brief version of the difficulties in emotion regulation scale (DERS-16; Bjureberg et al,. 2016) | Change in total score from baseline to 3-months post treatment (approximately 14-18 weeks).
  A 16-item self report measure of difficulties in emotion regulation. Total scores on the DERS-16 can range from 16 to 80, with higher scores reflecting greater levels of emotion dysregulation.
Work and Social Adjustment Scale (WSAS; Mundt et al., 2002) | Change in total score from baseline to 3-months post treatment (approximately 14-18 weeks).
  A 5-item self-report measure of work and social functioning and impact of symptoms. Total scores range from 0-40 with higher scores indicating greater impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Prevail Health Inc., Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McLean CP, Malek N, Straud CL. A pilot randomized controlled trial of online written exposure therapy delivered by peer coaches to veterans with posttraumatic stress disorder. J Trauma Stress. 2024 Jun;37(3):471-482. doi: 10.1002/jts.23020. Epub 2024 Feb 13. PMID 38348490